CLINICAL TRIAL: NCT03578315
Title: Advanced Harmonic Generation Microscopy for Treatment Assessment of Cutaneous Pigmentary Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201612113DINC
Record Dates: First submitted 2018-06-10; First posted 2018-07-06 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-06

CONDITIONS: Solar Lentigo; Nevus Zygomaticus
Keywords: Solar Lentigo; Nevus Zygomaticus; Harmonic Generation Microscopy; In Vivo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solar lentigo (Experimental): 25 Patients with Solar lentigo
  Interventions: Device: HGM
- Nevus zygomaticus (Experimental): 25 Patients with Nevus zygomaticus
  Interventions: Device: HGM

INTERVENTIONS:
Device: HGM — To Study the Efficacy and safety of QSRL and PSNYL in the Treatment of target: A nonrandomized, controlled, split-face comparative study

SUMMARY:
In this study, the investigators demonstrated that in vivo THG microscopy can differentiate Solar lentigos (SL), Nevus zygomaticus(NZ) and normal skin based on the optical nature of melanin. This THG-based procedure provides a valuable tool for noninvasive determination of third-order nonlinear susceptibility of melanin within the skin. It can also provide real-time histopathology information for treatment follow-up, without performing an invasive skin biopsy.

DETAILED DESCRIPTION:
A nonrandomized, controlled, split-face comparative study was conducted to compare the efficacy and safety between quality-switched ruby laser (QSRL) and 532-nm picosecond Nd:YAG laser (532-PSNYL for SL, 1064-PSNYL for NZ) in the treatment of solar lentigo clinically and histologically by harmonic generation microscopy (HGM). After baseline photography and in vivo harmonic generation microscopy (HGM) imaging, QSRL and 532-PSNYL or 1064-PSNYL therapy for solar lentigos and nevus zygomaticus on the left and right side of the face, respectively, were performed for each subject. The subjects underwent follow-up assessment at weeks 3 and 6.

Statistical analysis: All data gathered went through decoding and were analyzed by blinded evaluators using SPSS software (version 20.0; IBM, Armonk, NY). All tests were two-sided. A P value of < .05 was considered to be statistically significant.

ELIGIBILITY:
1. Main inclusion criteria:

1. Subjects are aged 20 to 85 years at Screening, and can be either sex.
2. Subjects are Fitzpatrick skin type III or IV.
3. Subjects must have been diagnosed to have solar lentigos or nevus zygomaticus, which are larger than 4 mm in diameter on both sides of the face.

2. Main exclusion criteria:

1. Subjects have previous treatments on the solar lentigos or nevus zygomaticus.
2. Subjects have a history of adverse reaction to laser treatments, including allergy to topical anesthesia application.
3. Subjects have a history of chronic inflammatory disorder such as atopic dermatitis on the face.
4. Subjects are pregnant or breast feeding.
5. Subjects have frequent sun exposure (≥4 hours per day).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
25 participants with Solar Lentigo and 25 participants with Nevus zygomaticus as assessed by clinical photographs | 6 months
  The primary endpoint is the improvement of target at week 6 scored with a 7-grade. physician global assessment

SECONDARY OUTCOMES:
25 participants with Solar Lentigo and 25 participants with Nevus zygomaticus as assessed by Harmonic Generation Microscopy. | 1-2 hours per case
  The HGM system will be combined to provide the noninvasive microscopic images in SL and NZ sites during each follow-up for pathological diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hua Liao, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan